CLINICAL TRIAL: NCT03310294
Title: A Randomized, Double Blind, Placebo-controlled Multicenter Clinical Study to Evaluate the Effect of a Combination of Probiotics and Prebiotics in Subjects With Recurrent Herpes Labialis
Brief Title: Immune Evidence to the Consumption of Lactobacillus GG and FOS Consumption in Patients With Herpes Labialis
Acronym: EVIM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-CLI-GRA-02
Record Dates: First submitted 2017-10-04; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Herpes Labialis
Keywords: Lactobacillus; Herpes Labial; Immune repsonse
MeSH Terms: conditions — Herpes Labialis | interventions — Prebiotics; Probiotics

STUDY DESIGN:
Intervention Model Description: This is a phase IV, parallel, placebo-controlled, double-blind, multicenter, randomized study to evaluate the effect of a combination of probiotics and prebiotics in subjects with recurrent Herpes labialis.
  This specific design has been chosen as the most suitable to achieve the objectives of the trial, mainly the demonstration of the clinical efficacy of the combination of probiotics and prebiotics in subjects with recurrent Herpes labialis in terms of reduction of the number of HL recurrences at day 49 vs baseline.
Who Masked: Participant, Investigator
Masking Description: As a double blind study neither the researchers nor the participants knew which treatment each participant received. The treatment was randomly allocated to the subjects according to the procedure for treatment assignment described above.
  To maintain the blind (see also paragraph 4.4.1) no differences between the active treatment and the placebo were evident on the package, and the carton boxes containing the study products were identified by a number corresponding to the randomization (the products will be labelled with a batch number, Investigator/center, subject ID number and expiry date).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): one bottle of placebo (minidrink fermented with low-fat milk but without Lactobacillus rhamnosus and without FOS, and without viable bacteria 90 grams)
  Interventions: Dietary Supplement: Placebo
- Prebiotics and Probiotics (Active Comparator): one bottle of the study product (minidrink with fermented low-fat milk added with Lactobacillus rhamnosus (Lactobacillus rhamnosus) and fructooligosaccharides (FOS), 90 grams)
  Interventions: Dietary Supplement: Prebiotics and Probiotics

INTERVENTIONS:
Dietary Supplement: Placebo — one bottle of placebo (minidrink fermented with low-fat milk but without Lactobacillus rhamnosus and without FOS, and without viable bacteria 90 grams)per day at breakfast until the end of the study (V5, day 140). At each visit, subjects were dispensed a sufficient amount of minidrinks until the next visit.
  Arms: placebo
Dietary Supplement: Prebiotics and Probiotics — one bottle of the study product (minidrink with fermented low-fat milk added with Lactobacillus rhamnosus (Lactobacillus rhamnosus) and fructooligosaccharides (FOS),per day at breakfast until the end of the study (V5, day 140). At each visit, subjects were dispensed a sufficient amount of minidrinks until the next visit.
  Arms: Prebiotics and Probiotics

SUMMARY:
Herpes labialis (HL) is the result of the presence of a virus called HSV-1 and is a common disease. Because of its visibility due to cold sores it has a serious impact on social life. Until now there is no effective treatment to prevent virus outbreaks. However, prebiotics and probiotics have both been shown to have a favorable and supportive effect on the immune system in different health conditions such as influenza, atopic dermatitis and diarrhea, so it is possible that they are able to have a favourable effect also on HL.

A recently completed pilot clinical trial (Protocol Number 08-SBUS-2-GRA-01, EVIM-1) was completed using a fermented milk (minidrink) containing a combination of L. rhamnosus and FOS; it showed promising results in the reduction of HL recurrences in a population of 78 subjects with HSV-1. The study investigated the effect of pre- or probiotics or a combination of the two on the recurrence of HL lesions as well as on the immune system in general, showing that the consumption of a minidrink containing the probiotic L. rhamnosus or a minidrink containing a combination of L. rhamnosus and FOS reduced the occurrence and the incidence of recurrent HL lesions.

Aim of this study: corroborate whether the consumption of a minidrink containing a combination of L. rhamnosus and FOS results in less recurrence and a better progression of HL lesion, in a larger population. In addition, the response of the consumption of the minidrink on the QoL and the response on immunity specific biomarkers were evaluated.

Design: 152 patients were eligible to participate in the study and after a run-in period of two weeks consuming a placebo minidrink were randomized to one of the two experimental study groups: placebo minidrink (n=79) and a minidrink containing a combination of a pre- and probiotic (n=78). These minidrinks were consumed until the end of the study (day 140). At day 33 of the study the lip most prone to the development of a lesion was stimulated with UVB to provoke a lesion. During the entire study period subjects were checked for any clinical signs of a lesion, completed a self-assessment regarding the lesion and a QoL questionnaire at baseline (day 14), at day 49 and the end of the study (day 140). In addition, a blood sample was collected at baseline, at day 49 and at the end of the study to be analyzed for HSV-specific antibody concentrations , to check immune system specific functions.

DETAILED DESCRIPTION:
Background: Herpes labialis is the result of the presence of HSV-1 and is a common disease. Because of its visibility it has a serious impact on social life. Until now there is no effective treatment to prevent virus outbreaks. However, prebiotics and probiotics have both been shown to have a favorable and supportive effect on the immune system in different health conditions such as influenza, atopic dermatitis and diarrhea.

A recently completed pilot clinical trial (Protocol Number 08-SBUS-2-GRA-01, EVIM-1) parallel groups, placebo controlled, triple blind, single center, randomized study, with a fermented milk (minidrink) containing a combination of L. rhamnosus and FOS showed promising results in the reduction of HL recurrences in a population of 78 subjects with HSV-1; the study investigated the effect of pre- or probiotics or a combination of the two on the recurrence of HL lesions as well as on the immune system in general, showing that the consumption of a minidrink containing the probiotic L. rhamnosus or a minidrink containing a combination of L. rhamnosus and FOS reduced the occurrence and the incidence of recurrent HL lesions.

Aim of the study: corroborate whether the consumption of a minidrink containing a combination of L. rhamnosus and FOS results in less recurrence and a better progression of HL lesion, in a larger population. In addition, the response of the consumption of the minidrink on the QoL and the response on immunity specific biomarkers were evaluated.

Design: 152 patients were eligible to participate in the study and after a run-in period of two weeks consuming a placebo minidrink were randomized to one of the two experimental study groups: placebo minidrink (n=79) and a minidrink containing a combination of a pre- and probiotic (n=78). These minidrinks were consumed until the end of the study (day 140). At day 33 of the study the lip most prone to the development of a lesion was stimulated with UVB to provoke a lesion. During the entire study period subjects were checked for any clinical signs of a lesion, completed a self-assessment regarding the lesion and a QoL questionnaire at baseline (day 14), at day 49 and the end of the study (day 140). In addition, a blood sample was collected at baseline, at day 49 and at the end of the study to be analyzed for HSV-specific antibody concentrations (circulating concentrations of IgG1 and IgG3 (Th1) and IgG4 (Th2), NK activity, CXCL10 analyzed by ELISA at days 14, 49 and 140).

as regards the primary endpoint results have shown that there was a significant decrease (54.3%) in the recurrences of Herpes labialis lesions, post UV stimulation, at day 49 (V4) compared to placebo in the PP population with consumption of the study product minidrink with fermented low fat milk added with Lactobacillus rhamnosus and FOS. Considering the secondary endpoints in the PP population, considering the number of subjects who presented lesions between V0 and V5, the number of lesions is reduced significantly (both statistically and clinically) in the treatment group compared to the placebo group. There was a decrease in the lesion size in the treatment group when compared to placebo although the statistical significance is marginal. As regards 'Subjective assessment of pain', evaluated by means of a VAS scale, significant pain reduction was found in the treatment group compared to the placebo group. As regards immunological parameters was shown an increase in CXCL10 at V4 in the study group compared to the placebo group. As regards IgG1, IgG3 and IgG4 (V0, V4 and V5) although substantial increases were registered for some of these parameters, these were not sufficient to describe a definite trend. The natural killer (NK) cell activity did not show significant difference in their functional activity in the treatment group as compared to the placebo group.

It has been verified through quality of life questionnaire (SF-36 questionnaire) that treatment improved Mental Health in the treatment group (Nervous, Peaceful, Happy, Down in Dumps, Sad) compared to the placebo group and clinical significance was found at V4 and V5. General Health and Vitality has been improved at V4 and V5.

For each trial participant the adverse events/serious adverse events occurrences and a brief clinical examination were assessed. No special or unusual features of the safety evaluations were found.

ELIGIBILITY:
Inclusion Criteria:

* Healthy free-living men and women aged 18 to 65 years-old.
* History of recurrent HL (2 - 4 episodes) after exposure to sunlight in the previous 12 months.
* Fitzpatrick skin type 1 to 4 (appendix 1 of the study protocol).
* No presence of HL lesions at time of recruitment, including baseline.
* Agreement to adhere to the prescribed list of dietary recommendations provided at the start of the study (appendix 3 of the study protocol).
* Women of child-bearing potential are required to use adequate birth protection during the study.
* Sign and date the ICF to and to comply with study procedures

Exclusion Criteria:

* Presence of acute/terminal disease.
* Intolerance for milk protein or lactose.
* Treatment with acyclovir or other medication believed to interfere with immune responses at the time of the study.
* Participation in any herpes UV reactivation study within the previous three months.
* Pregnancy or lactation.
* Any condition (e.g. schizophrenia, psychosis, major depression or mental deficiency) or major co-morbidity that the study investigator thinks might compromise the person's ability to comply with the requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2010-09-14 (Actual); Primary Completion 2011-05-05 (Actual); Study Completion 2011-08-01 (Actual)

PRIMARY OUTCOMES:
reduction of HL recurrence. | Day 49
  to evaluate the coadjuvant effect of the combination of prebiotic and probiotic mix in the reduction of the number of HL recurrences at day 49 vs baseline.

SECONDARY OUTCOMES:
reduction of HL recurrence. | day 14
  to evaluate the coadjuvant effect of the combination of prebiotic and probiotic mix in the reduction of the number of HL recurrences at day 49 vs baseline.
reduction of HL recurrence. | day 140
  to evaluate the coadjuvant effect of the combination of prebiotic and probiotic mix in the reduction of the number of HL recurrences at day 49 vs baseline.
change IGS markers concentration | day 14
  Evaluate the effect of the combination of prebiotic and probiotic mix on specific IGs markers;
change IGS markers concentration | day 49
  Evaluate the effect of the combination of prebiotic and probiotic mix on specific IGs markers;
change IGS markers concentration | day 140
  Evaluate the effect of the combination of prebiotic and probiotic mix on specific IGs markers;
time to healing | Day 14
  Evaluate the coadjuvant effect of the combination of prebiotic and probiotic mix in the time to healing, defined as either loss of the hard crust or return to normal skin (measured in days);
time to healing | Day 49
  Evaluate the coadjuvant effect of the combination of prebiotic and probiotic mix in the time to healing, defined as either loss of the hard crust or return to normal skin (measured in days);
time to healing | Day 140
  Evaluate the coadjuvant effect of the combination of prebiotic and probiotic mix in the time to healing, defined as either loss of the hard crust or return to normal skin (measured in days);
lesion size | Day 14
  Evaluate measurement of lesion size as a product of the length and the width of the lesion development (measured in mm2) by classification of lesion stage
lesion size | Day 49
  Evaluate measurement of lesion size as a product of the length and the width of the lesion development (measured in mm2) by classification of lesion stage
lesion size | Day 140
  Evaluate measurement of lesion size as a product of the length and the width of the lesion development (measured in mm2) by classification of lesion stage
SF-36 | Day 14
  Evaluate quality of life by means of SF-36 questionnaire
SF-36 | Day 49
  Evaluate quality of life by means of SF-36 questionnaire
SF-36 | Day 140
  Evaluate quality of life by means of SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michelangelo La Placa, master, Principal Investigator — Dipartimento di Medicina Interna, dell'Invecchiamento e Malattie Nefrologiche Università degli Studi di Bologna